CLINICAL TRIAL: NCT03187210
Title: Brentuximab Vedotin and BeEAM High-dose Chemotherapy (B-BeEAM) With Autologous Stem Cell Transplantation for CD30+ Lymphomas, a Phase I/II Study
Brief Title: Brentuximab Vedotin and BeEAM High-dose Chemotherapy in Lymphomas
Acronym: BAL
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Mundipharma Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAL-Trial
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma
Keywords: CD30+ Lymphoma; ASCT; Brentuximab Vedotin
MeSH Terms: conditions — Lymphoma | interventions — Brentuximab Vedotin

STUDY DESIGN:
Intervention Model Description: The BAL trial consists in two parts:
  * single arm prospective phase I part;
  * randomized two-arm open-label prospective phase II part.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dosis finding (Phase I) (Experimental): Brentuximab Vedotin at day -8 together with standard BeEAM (Bendamustine, Cytarabine, Etoposide and Melphalan) chemotherapy at days -7 to -1 followed by reinfusion of autologous stem cells at day 0
  Interventions: Drug: Brentuximab Vedotin; Drug: BeEAM Regimen
- Arm A (Phase II) (Active Comparator): BeEAM Regimen:
  Bendamustine intravenously once daily on days -7 and -6 at 200 mg/m2/day; Cytarabine (ARA-C) 400 mg/m2/day intravenously once daily from day -5 to day-2; Etoposide 200 mg/m2/day intravenously once daily from day -5 to day -2; and Melphalan 140 mg/m2/day intravenously once on day -1, followed by reinfusion of autologous stem cells at day 0
  Interventions: Drug: BeEAM Regimen
- Arm B (Phase II) (Experimental): Brentuximab Vedotin 1.8 mg/kg at day -8 together with standard BeEAM chemotherapy at days -7 to -1
  BeEAM Regimen:
  Bendamustine intravenously once daily on days -7 and -6 at 200 mg/m2/day; Cytarabine (ARA-C) 400 mg/m2/day intravenously once daily from day -5 to day-2; etoposide 200 mg/m2/day intravenously once daily from day -5 to day -2; and Melphalan 140 mg/m2/day intravenously once on day -1, followed by reinfusion of autologous stem cells at day 0
  Interventions: Drug: Brentuximab Vedotin; Drug: BeEAM Regimen

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab Vedotin at day -8 together with standard BeEAM chemotherapy at days -7 to -1 followed by ASCT on day 0
  Arms: Arm B (Phase II); Dosis finding (Phase I)
Drug: BeEAM Regimen — standard BeEAM chemotherapy at days -7 to -1 followed by ASCT on day 0

SUMMARY:
The trial assess the maximum tolerated dose of a single-dose of Brentuximab Vedotin added to standard BeEAM chemotherapy (comprising Bendamustin, Etoposide, Cyclophosphamide and Melphalan) before autologous stem cell transplantation in CD30+ malignant lymphomas.

DETAILED DESCRIPTION:
Background and Rationale:

CD30+ lymphomas typically comprise Hodgkin lymphomas and a variety of T-cell non-Hodgkin lymphoma (T-NHL) entities including angioimmunoblastic T-cell lymphomas (AITL), anaplastic ALK+ large-cell T-cell lymphomas (ALCL), Sézary-syndrome, peripheral T-NHL NOS and other rare malignant T-cell lymphoma types.

The prognosis of patients with Hodgkin lymphoma (HL) is excellent for the majority of these usually young patients; however, HL patients relapsing after autologous stem-cell transplantation (ASCT) have a rather poor outcome, with approximately only up to 20% of the patients surviving longer than 5 years. For those in advanced stage Hodgkin's lymphoma multiple first-line and second-line treatments, including the combination of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) - internationally, the most widely used regimen in Hodgkin's lymphoma - is expected to cure about 70-80% of patients. However, in addition to treatment failures noted for ABVD, the regimen is often associated with unpredictable bleomycin-induced lung related toxic effects that can be life-threatening. Although High Dose Chemotherapy (HDCT) with ASCT is a curative strategy for some patients with relapsing Hodgkin lymphomas, relapse or progression after ASCT is a major limitation of this procedure. For these reason, the outcome of Hodgkin lymphoma patients relapsing after ASCT is poor, and novel concepts for such patients is an unmet clinical need.

CD30+ T-NHL generally have a limited prognosis, with a minority of patients being cured after specific lymphoma treatment. The incorporation of consolidating high-dose chemotherapy with autologous stem cell transplantation for young fit patients within the first-line treatment algorithms has improved the prognosis of such patients to some extent. However, the majority of such patients still ultimately die of their disease. Again, improvement of lymphoma treatment is an urgent requirement for these patients.

Brentuximab Vedotin (BV; Adcetris®) is an antibody-drug conjugate and is licensed in Switzerland and the European Medicine Agency region for the single-agent treatment of relapsed and refractory Hodgkin lymphoma or for relapsed and refractory anaplastic T-cell lymphoma.

BeEAM high-dose chemotherapy (comprising Bendamustin, Etoposide, Cyclophosphamide and Melphalan) is the standard conditioning regimen before ASCT for lymphoma patients.

In this trial BV will be used together with BeEAM high-dose chemotherapy according to its conventional schedule in CD30+ lymphomas as conditioning regimen before ASCT.

Objective:

Phase I: The primary objective of the trial is to assess the maximum tolerated dose of a single-dose of Brentuximab Vedotin added to standard BeEAM chemotherapy before autologous stem cell transplantation in CD30+ malignant lymphomas.

Phase II: The main objective of the trial is to assess differences in disease-free survival between CD30+ lymphoma patients treated with the standard BeEAM high-dose chemotherapy versus Brentuximab Vedotin together with BeEAM (B-BeEAM) high-dose chemotherapy. We aim to demonstrate an improvement by 20% of the rate of disease-free survival 1 year after ASCT (DFS1) from 70% in patients treated with BeEAM alone to 90% in patients treated with the combination of B-BeEAM.

Study Duration:

Phase I part was planned to last from 3 to 18 months (permitting the enrolment of minimum of 6 patients). The Phase I has been stopped after the RP2D (1.8mg/kg/day) was established with enrolment of 12 patient in 24 months. The Phase II will stop after the inclusion of 42 evaluable patients.

All patients will be followed up for up to 12 months after end of treatment..

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP or ISO EN 14155 (as far as applicable) as well as all national legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Eligible are all CD30+ malignant lymphoma, meaning lymphoma subtypes such as Hodgkin lymphomas, angioimmunoblastic T-cell lymphomas (AITL), anaplastic ALK+ T-cell lymphomas, Sézary-syndrome, but also all other malignant CD30+ lymphoma types.
* Patients must be in first or second remission or second chemosensitive relapse and patients must be planned to undergo subsequent consolidation with standard high-dose chemotherapy with autologous stem cell transplantation.
* Patients must be aged 18-75 years, and must have given voluntary written informed consent.
* Negative pregnancy test (urine or serum) within 14 days prior to registration for all women of childbearing potential. Patients of childbearing potential must implement two effective contraceptive measures (hormonal treatment p.o. or i.m., intra uterine surgical devices, or latex condoms) to avoid pregnancy from the time of signing informed consent and for additional 12 months. No pregnant or lactating patients are allowed.
* Male patients, even if surgically sterilized, (i.e., status post vasectomy) agree to practice effective barrier contraception during the entire study period and through 12 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
* Absolute neutrophil count ≥ 1,500/µL unless there is known hematologic/solid tumor marrow involvement.
* Platelet count ≥ 75,000/ µL unless there is known marrow involvement of the disease.
* Total bilirubin must be < 1.5 x the upper limit of the normal (ULN) unless the elevation is known to be due to Gilbert syndrome.
* ALT or AST must be < 3 x the upper limit of the normal range. AST and ALT may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of hematologic/solid tumor in liver.
* Serum creatinine must be < 2.0 mg/dL and/or calculated creatinine clearance > 40 mL/minute (Cockcroft-Gault).
* Hemoglobin must be ≥ 8g/dL.

Exclusion Criteria:

* Patients considered to be not fit for autologous stem cell transplantation (ASCT).
* Patients with other serious medical condition that interfere with the completion of treatment according to this protocol or that would impair tolerance to therapy or prolong hematological recovery. Patients with seropositivity for HIV or for Hepatitis B and C are not excluded from this study if they are otherwise considered fit for ASCT.
* Symptomatic neurologic disease compromising normal activities of daily living or requiring medications. Any sensory or motor peripheral neuropathy greater than or equal to Grade 2.
* Known history of any of the following cardiovascular conditions: Myocardial infarction within 2 years of registration, New York Heart Association (NYHA) Class III or IV heart failure (See Appendix 5). Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities, Recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction <50%.
* Patients that have not completed any prior treatment chemotherapy and/or other investigational agents within at least 5 half-lives of last dose of that prior treatment. Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of Brentuximab Vedotin.
* Acute uncontrolled infection.
* Relevant co-existing disease excluding a treatment according to protocol.
* Concurrent malignant disease with the exception of basalioma/spinalioma of the skin, early-stage cervix carcinoma, or early-stage prostate cancer. • Previous treatment for other malignancies (not listed above) must have been terminated at least 24 months before registration and no evidence of active disease must be documented since then.
* Lack of patient cooperation to allow study treatment as outlined in this protocol.
* Pregnant or lactating female patients.
* Major coagulopathy or bleeding disorder.
* Major surgery less than 30 days before start of treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose finding | 30 days
  To identify the maximum tolerated dose of Brentuximab Vedotin added to standard BeEAM high-dose chemotherapy testing three dose levels.
Phase 2: Disease free survival at 12 months | 12 months
  Number of patients with disease-free survival 12 months after ASCT (DFS1) between CD30+ lymphoma patients treated with the standard BeEAM high-dose chemotherapy versus brentuximab together with BeEAM (B-BeEAM) high-dose chemotherapy. A clinically meaningful increase of the efficacy of the combination therapy (B-BeEAM) is defined in this study as an increase of the rate of disease free survival (DFS1) one year after ASCT from 70% with BeEAM alone to ≥ 90% with the combination of Brentuximab Vedotin and BeEAM.

SECONDARY OUTCOMES:
Phase 1: Disease-free survival | 12 months
  Number of patients with disease-free survival 12 months after ASCT
Phase I and II: Overall survival | 12 months
  Number of patient alive after 12 months
Phase II: Overall response rate | 12 months
  Number of patients experiencing complete or partial remission
Phase I and II: Adverse Events | 12 months
  Number of patient experiencing toxicity (Adverse events)
Phase I and II: Engraftment and hematologic recovery | 30 days
  Number of days until neutrophils recovery 0.5 G/L (from day - 8)
Phase I and II: Infectious complications | 12 months
  Number of patients experiencing infectious complications
Phase I and II: Overall response rate | 12 months
  Number of patients experiencing complete or partial remission

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pabst, MD, Study Chair — Department of Medical Oncology, University Hospital Bern
Locations (1):
- Department for Medical Oncology University Hospital/Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Rausch C, Bacher U, Rabaglio M, Vorburger C, Klingenberg A, Banz Y, Daskalakis M, Pabst T. Randomized Phase II Study of Brentuximab-Vedotin With High-Dose Chemotherapy in CD30 Positive Lymphoma. Hematol Oncol. 2025 Nov;43(6):e70143. doi: 10.1002/hon.70143. PMID 41117344